CLINICAL TRIAL: NCT05462262
Title: Effects of Intensive Lipid-lowering on Coronary Atherosclerotic Plaque Phenotype and Major Adverse Cardiovascular Events in Adults With Low to Intermediate 10-year ASCVD Risk: a Prospective, Randomized, Open-label, Blinded Endpoint Analysis(PROBE)
Brief Title: Intensive Lipid-lowering for Plaque and Major Adverse Cardiovascular Events in Low to Intermediate 10-year ASCVD Risk Population
Acronym: ILLUMINATION
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Bin Lu, Principle Investigator of National Center for Cardiovascular Diseases and National Clinical Research Center of Cardiovascular Diseases, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-CXGC03-3
Record Dates: First submitted 2022-07-07; First posted 2022-07-18 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease Progression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: blinded endpoint
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intensive lipid-lowering group (Experimental): Goal for LDL-C <1.8 mmol/L or ≥50% reduction from baseline.
  Interventions: Drug: Intensive lipid-lowering control
- moderate-intensity lipid-lowering group (Active Comparator): Goal for LDL-C <2.6 mmol/L or 30%-50% reduction from baseline.
  Interventions: Drug: Moderate-intensity lipid-lowering control

INTERVENTIONS:
Drug: Intensive lipid-lowering control — The initial recommended therapy is 10-20mg atorvastatin plus Ezetimibe, and the type and dosage of drugs can be adjusted according to the situation.
  Other Names: Lower goal for reducing LDL-C
  Arms: intensive lipid-lowering group
Drug: Moderate-intensity lipid-lowering control — The initial recommended therapy is 10-20mg atorvastatin, and the type and dosage of drugs can be adjusted according to the situation.
  Other Names: Standard goal for reducing LDL-C
  Arms: moderate-intensity lipid-lowering group

SUMMARY:
Current guidelines recommend moderate-intensity lipid-lowering therapy (goal for LDL-C <2.6 mmol/L or 30%-50% reduction from baseline) for patients with intermediate 10-year ASCVD risk. In these patients, early coronary atherosclerotic plaques detected by coronary CT angiography are common, but further interventions are lacking. This study aims to analyze whether intensive lipid-lowering therapy (goal for LDL-C <1.8 mmol/L or ≥50% reduction from baseline) could delay the progression of coronary atherosclerotic lesions and reduce the adverse cardiovascular events in these target patients.

DETAILED DESCRIPTION:
Both American (2019 ACC/AHA Guideline on the Primary Prevention of Cardiovascular Disease) and European (2019 ESC/EAS Guidelines for the management of dyslipidemias) guidelines currently recommended moderate-intensity lipid-lowering (goal for LDL-C <2.6 mmol/L or 30%-50% reduction from baseline) for primary prevention in the population at intermediate (or borderline) 10-year ASCVD risk, but the residual risk in this group of the population remains to be explored, especially in a subset with only nonobstructive atherosclerotic plaques detected by CCTA, for whom further risk stratification and precise interventions for primary prevention are lacking.

CCTA could show accurate images of patients' early coronary atherosclerotic lesions and provides a wealth of image-based anatomical and functional information including plaque burden (total plaque volume, calcification score, segment involvement score, etc.), plaque composition, high-risk plaque characteristics, luminal stenosis, and CT-FFR. With this complete imaging information on CCTA, there is an urgent need to investigate primary prevention strategies and the evidence-based rationale for performing precise risk stratification in low to intermediate-risk populations with nonobstructive coronary atherosclerotic lesions using CCTA.

A prospective, randomized, open-label, blinded endpoint analysis (PROBE) will be conducted in the population at clinical low to intermediate 10-year ASCVD risk with nonobstructive coronary atherosclerotic lesions, predominantly non-calcified plaques detected by CCTA. The purpose of this study is to demonstrate that intensive lipid-lowering could slow down plaque progression and reduce the incidence of MACE in the target population, which provides an evidence-based rationale for further risk re-stratification. Enrolled people will be randomized into the intervention group (goal for LDL-C <1.8 mmol/L or ≥50% reduction from baseline) and the control group (goal for LDL-C <2.6 mmol/L or 30%-50% reduction from baseline).

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-75 years
2. Low to Intermediate 10-year atherosclerotic cardiovascular disease (ASCVD) risk using pooled cohort equations (PCE).
3. Coronary CT angiography shows atherosclerotic plaque in the main coronary vessels (>2mm diameter) with luminal stenosis <70%

Exclusion Criteria:

1. Combination with serious cardiovascular diseases, including

   1. Heart failure (ejection fraction <30%)
   2. Arrhythmias (persistent atrial flutter/atrial fibrillation, second-degree or third-degree atrioventricular block)
   3. Hemodynamically important valvular disease
   4. Hemodynamically important congenital heart disease
   5. Stroke
2. Myocardial infarction, coronary revascularization, or severe/unstable angina before or within 1 month of screening
3. Active liver disease or hepatic dysfunction (defined as alanine aminotransferase or aspartate aminotransferase> 3 times the upper limit of normal)
4. Unexplained creatine phosphokinase> 6 times the upper limit of normal
5. Nephrotic syndrome
6. Diabetes mellitus
7. Uncontrollable hypertension
8. Uncontrollable hypothyroidism
9. Hypersensitivity to statins
10. Any planned surgical procedure for the treatment of atherosclerosis
11. Gastrointestinal diseases affecting drug absorption or history of gastrointestinal surgery
12. Survival-limiting diseases
13. Concurrent long-term immunosuppressive therapy
14. Participation in another clinical trial concurrently or within 30 days before screening
15. Pregnant or breastfeeding
16. Other unsuitable situations deemed by physicians

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2900 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | Within 3 years after the enrollment
  Composite of all-cause death, non-fatal MI, non-fatal stroke, any revascularization, and hospitalization for angina

SECONDARY OUTCOMES:
Change in coronary total plaque volume(mm³) on CCTA | Within 3 years after the enrollment
  Total plaque volume(mm³) is defined as the sum of all plaque volumes for coronary arteries.
Change in coronary plaque burden(%) on CCTA | Within 3 years after the enrollment
  Plaque burden(%)=(plaque area/vessel area)×100%
Changes in coronary plaque compositions(mm³, %) on CCTA | Within 3 years after the enrollment
  Plaque compositions include lipid(<30 HU), fibrous(30-150HU), and calcified plaque(>350HU).
Changes in coronary high-risk plaque characteristics on CCTA | Within 3 years after the enrollment
  High-risk plaque characteristics are defined as positive remodeling(remodeling index, >1.1), low CT attenuation (mean CT number <30 HU), spotty calcification(punctate calcium within a plaque measuring less than 3 mm in all dimensions), or napkin-ring sign (a ringlike peripheral higher attenuation with central low CT attenuation).
Change in coronary artery calcium score (CACS) on CT | Within 3 years after the enrollment
  CACS is a quantification of all coronary calcification by the scoring algorithm proposed by Agatston et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mach F, Baigent C, Catapano AL, Koskinas KC, Casula M, Badimon L, Chapman MJ, De Backer GG, Delgado V, Ference BA, Graham IM, Halliday A, Landmesser U, Mihaylova B, Pedersen TR, Riccardi G, Richter DJ, Sabatine MS, Taskinen MR, Tokgozoglu L, Wiklund O; ESC Scientific Document Group. 2019 ESC/EAS Guidelines for the management of dyslipidaemias: lipid modification to reduce cardiovascular risk. Eur Heart J. 2020 Jan 1;41(1):111-188. doi: 10.1093/eurheartj/ehz455. No abstract available. PMID 31504418
- [Background] Arnett DK, Blumenthal RS, Albert MA, Buroker AB, Goldberger ZD, Hahn EJ, Himmelfarb CD, Khera A, Lloyd-Jones D, McEvoy JW, Michos ED, Miedema MD, Munoz D, Smith SC Jr, Virani SS, Williams KA Sr, Yeboah J, Ziaeian B. 2019 ACC/AHA Guideline on the Primary Prevention of Cardiovascular Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Sep 10;140(11):e596-e646. doi: 10.1161/CIR.0000000000000678. Epub 2019 Mar 17. No abstract available. PMID 30879355
- [Background] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Jun 18;139(25):e1082-e1143. doi: 10.1161/CIR.0000000000000625. Epub 2018 Nov 10. PMID 30586774
- [Derived] Zheng J, Hou Z, Yuan J, Zhao X, Wang Y, Li J, Zhang W, Dou K, Lu B. Effects of intensive lipid lowering compared with moderate-intensity lipid lowering on coronary atherosclerotic plaque phenotype and major adverse cardiovascular events in adults with low to intermediate 10-year ASCVD risk (ILLUMINATION study): protocol for a multicentre, open-label, blinded-endpoint, randomised controlled trial. BMJ Open. 2023 Jun 5;13(6):e070832. doi: 10.1136/bmjopen-2022-070832. PMID 37277217
- See also: China-PAR 10-year ASCVD risk model — https://www.cvdrisk.com.cn/ASCVD/Eval